CLINICAL TRIAL: NCT01509755
Title: Dose-response Relationship of Five Dose Levels of NNC90-1170 and Placebo on Glycaemic Control in Type 2 Diabetic Patients Compared to OHA Treatment. A 12-week Multi-centre, Double-blind, Randomised, Parallel Group Trial With an Open Labelled OHA Arm
Brief Title: Comparison of Liraglutide and Glimepiride on Blood Sugar Control in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN2211-1310
Record Dates: First submitted 2012-01-06; First posted 2012-01-13 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- 0.045 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.225 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.45 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.60 mg (Experimental)
  Interventions: Drug: liraglutide
- 0.75 mg (Experimental)
  Interventions: Drug: liraglutide
- Glim (Active Comparator)
  Interventions: Drug: placebo; Drug: glimepiride

INTERVENTIONS:
Drug: placebo — Once daily injection, under the skin (s.c.) for 12 weeks
  Arms: Glim; Placebo
Drug: liraglutide — Once daily injection, under the skin (s.c.) for 12 weeks
  Other Names: NNC 90-1170
  Arms: 0.045 mg; 0.225 mg; 0.45 mg; 0.60 mg; 0.75 mg
Drug: glimepiride — Tablets administered orally according to current treatment guidelines. Dose adjusted according to the glycaemic response
  Arms: Glim

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to establish the dose response relationship on glycaemic control of five dose levels of NNC90-1170.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* Duration of diabetes at least 3 months
* Both diet treated and patients in therapy with OHA (oral hypoglycemic agents)
* Body Mass Index maximum 40 kg/m^2
* HbA1c based on analysis from central laboratory: Between 7.5-10.0%, both inclusive, for diet treated, or maximum 9.0% for OHA treated

Exclusion Criteria:

* Liver or renal disease
* Cardiac problems
* Uncontrolled treated/untreated hypertension
* Proliferative retinopathy
* Recurrent severe hypoglycaemia as judged by the Investigator
* Known or suspected allergy to trial product or related products
* Use of any drug (except for OHAs) which in the Investigator's opinion could interfere with the blood glucose level

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2000-10; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

PRIMARY OUTCOMES:
HbA1c (glycosylated haemoglobin)

SECONDARY OUTCOMES:
Fasting plasma glucose
Fructosamine
7-point blood glucose profile
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), MD, Study Director — Novo Nordisk A/S
Locations (29):
- Denmark (6):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Kolding
  - Novo Nordisk Investigational Site, Køge
  - Novo Nordisk Investigational Site, Thisted
- Norway (4):
  - Novo Nordisk Investigational Site, Bekkestua
  - Novo Nordisk Investigational Site, Elverum
  - Novo Nordisk Investigational Site, Harstad
  - Novo Nordisk Investigational Site, Oslo
- Sweden (5):
  - Novo Nordisk Investigational Site, Gothenburg
  - Novo Nordisk Investigational Site, Grästorp
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Örebro
  - Novo Nordisk Investigational Site, Uppsala
- United Kingdom (14):
  - Novo Nordisk Investigational Site, Ayrsh
  - Novo Nordisk Investigational Site, Church Village
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Enfield
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Leicester
  - Novo Nordisk Investigational Site, Liverpool
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Nottingham
  - Novo Nordisk Investigational Site, Oxford
  - Novo Nordisk Investigational Site, Plymouth
  - Novo Nordisk Investigational Site, Rugby
  - Novo Nordisk Investigational Site, Sheffield
  - Novo Nordisk Investigational Site, Worksop

REFERENCES:
- [Result] Madsbad S, Schmitz O, Ranstam J, Jakobsen G, Matthews DR; NN2211-1310 International Study Group. Improved glycemic control with no weight increase in patients with type 2 diabetes after once-daily treatment with the long-acting glucagon-like peptide 1 analog liraglutide (NN2211): a 12-week, double-blind, randomized, controlled trial. Diabetes Care. 2004 Jun;27(6):1335-42. doi: 10.2337/diacare.27.6.1335. PMID 15161785
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com